CLINICAL TRIAL: NCT02347566
Title: The Efficacy of a Physical Activity Enhancing Programme Using Activity Monitors With Set Targets and Feedback for Enhancing Physical Activity Levels in Patients With COPD Attending Pulmonary Rehabilitation.
Brief Title: Physical Activity Enhancing Programme in COPD
Acronym: PAEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/0380
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Physical Activity; Accelerometer
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical activity enhancing programme (Experimental): Usual care + physical activity enhancing programme (PAEP) (Study group, [S]), which includes both pulmonary rehabilitation programme plus the PAEP using an activity monitor (DirectLife) with set targets of physical activity levels to stimulate and increase physical activity in daily life.
  Interventions: Behavioral: Physical activity enhancing programme
- Control (Other): Usual care (control, [C]) that includes only the pulmonary rehabilitation programme with the use of an activity monitor (DirectLife) in daily routine without any feedback or incentive to increase physical activity in daily life.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Physical activity enhancing programme — COPD patients performing pulmonary rehabilitation will wear the DirectLife activity monitor with set targets and feedback. They will have access to a web coaching programme. Their physical activity targets will be updated on a weekly basis in order to enhance their physical activity.
  Arms: Physical activity enhancing programme
Other: Usual care — COPD patients performing pulmonary rehabilitation will wear the DirectLife activity monitor without set targets and/or feedback. They will not have access to a web coaching programme.
  Arms: Control

SUMMARY:
Patients with Chronic Obstructive Pulmonary Disease are characterised by a sedentary lifestyle. This contributes to increase the number of hospitalizations and mortality. Changing this lifestyle is a major objective of the management of these patients. Pulmonary rehabilitation helps patients to increase their fitness, but modifying a longstanding sedentary habit is more difficult to achieve. This project aims at modifying patients' long term physical activity with a physical activity coaching programme. This will help patients to transform the benefits of pulmonary rehabilitation into a healthier active lifestyle and contribute to reduce hospitalizations, increase quality of life and survival.

DETAILED DESCRIPTION:
Study Design:

For logistical purposes, the study is divided into two work packages (WP): 1) Pilot study of DirectLife activity monitor in the daily routine of patients with COPD (WP1), which is a cross-sectional study; 2) Physical activity enhancing programme - main project (WP2), which is a randomized controlled trial. Both studies will be performed at Leith's Community Treatment Centre (LCTC) and its satellites (Midlothian Community Hospital (Bonnyrigg) & St Johns Hospital (Livingston) - Edinburgh). Only patients with COPD referred to pulmonary rehabilitation at LCTC and its satellites will be recruited for this study. The standard care treatment (exercise training) is exactly the same in all sites, and it is delivered by the same team of physiotherapists.At the satellite units it would still be the direct care that approach the participants. The recruiting procedure will be the same as that of the original study.

Written and signed consent will be taken prior to the inclusion of each patient. The study will explain the protocol and all the procedures they may undergo during study period before they sign the informed consent. With at least 24 hours in advance and before considering patients to take part in the study, we will send them the patient information sheet explaining the project and all the procedures involved.

WP1: This WP aims at establishing the best wearing position of the DirectLife activity monitor in 20 patients with COPD in their daily routine at home. As the DirectLife was only validated in healthy subjects, this is an important step to understand how this device works in daily routine, which is the best position to wear it, and also how feasible it is to use in patients with COPD.

This WP will be conducted prior to the beginning of WP2 and participants will sign a consent form to participate in the study. Twenty COPD patients will undertake the following assessments: pulmonary function (spirometry), exercise capacity (ISWT and ESWT), quality of life (CRQ), dyspnoea sensation (MRC scale) and physical activity in daily life.

Patients will wear simultaneously three different DirectLife devices in three different body places (on the hip, in the front pocket and on the neck) and a fourth physical activity monitor (Actigraph GT3x) which was recently shown as a valid and accurate device to measure daily PAL in patients with COPD.

Patients will wear all four activity monitors (three DirectLife and one Actigraph GT3x) simultaneously in their daily routine, for a period of at least 10 hours/day during the evaluation period of one week. After this monitoring period, they will answer a simple questionnaire about the feasibility of using DirectLife in day-to-day including questions such as: which position(s) they considered as the best position to wear DirectLife, how easy was to put it on and whether the use of DirectLife interfered or not in their daily routine. At the end of this WP we will be able to establish the best position to use the DirectLife and this position will be used in the WP2. If one site is not favoured over the others for monitor position, we will ask patients to wear DirectLife at the place they judge as the most comfortable. If DirectLife does not provides an accurate measurement of patients' physical activity, we will ask them to wear the device in the pocket (position that the manufacturer states it is the best to wear it).

WP2: This WP aims at comparing a PAEP added to pulmonary rehabilitation against usual care (pulmonary rehabilitation alone). Sixty-four patients with COPD will be randomized into two groups: Usual care (control, [C]) that includes only the pulmonary rehabilitation programme with the use of the DirectLife in daily routine without any feedback or incentive to increase PAL; or usual care + physical activity enhancing programme (PAEP) (Study group, [S]), which includes both pulmonary rehabilitation programme plus the PAEP using the DirectLife activity monitor with set targets of physical activity levels to stimulate and increase PADL. Both groups will perform the same pulmonary rehabilitation programme, composed by (in brief): resistance training of quadriceps femoris, biceps and triceps brachii; aerobic exercises in treadmill and cycle ergometer during 6-10 weeks.

All patients will be assessed before PR (Visit 1), and 3 months after the beginning of PR (Visit 2). Patients will be followed up by 3 months after visit 2 (Visit 3).

Assessment will include lung function (spirometry), exercise capacity, peripheral muscle strength, physical activity in daily life, quality of life, systemic inflammation, anxiety and depression, and dyspnoea sensation (see description below). In addition, patients will fill in a psychological survey on three occasions: visit 1, visit 2, and end of the study (visit 3).

For the follow-up phase, patients from both groups (S and C) will be invited to attend the same assessments performed in Visit 1 (excluding spirometry, ISWT and blood samples), three months after visit 2 (Visit 3) to assess the maintenance of the effects of the programme. This additional monitoring period is optional. Therefore patients can choose whether they want to keep helping us with the study or not. For this three months period, both groups will be wearing the DirectLife (without any feedback or incentive to increase physical activity) to monitor PAL over that period. Over this three months follow up period, patients will not receive any formal physical activity counseling/intervention, and they will be excluded from the analysis if they would be under any treatment that could influence their PAL (i.e., pulmonary rehabilitation).

In both groups, initial physical activity levels (PALi) will also be established by assessing PAL with the DirectLife activity monitor (DirectLife, Philips, The Netherlands) throughout a whole week. The physical activity data collected by the DirectLife activity monitor will be used to facilitate the behavioural intervention in the S group, but not as an outcome of PAL for which a different activity monitor (Actigraph GT3x) validated in COPD will be used. The DirectLife activity monitor is a lightweight and portable device that can be worn in three different places (necklace, on the pocket or on the hip) and provides as main variables the active time (minutes) and energy expenditure (calories). DirectLife tracks the body motion with its triaxial sensor. It also provides feedback to the patients on PAL performed since the beginning of the day; a series of indicator lights on the Activity Monitor shows the accumulated activity at any particular moment of each day. It also shows the daily target of physical activity levels making it easy for them to keep on track towards their goals. The aim of the study will be to achieve increments in 50% of the initial PAL at the end of the 12 weeks programme in the S group.

Exercise training programme

Both groups will perform a 6-10 weeks standard exercise training programme used in the UK, 1-2 times per week. Each training session will last 1 hour. As mentioned before, the exercise programme will include cycling; walking; and strength training for the quadriceps femoris, biceps, and triceps brachii muscle groups. The physiotherapist at LCTC and its satellites will increase the work rate or duration of the exercise programme every week guided by a pre-determined schedule and driven by the patient's perception of symptoms (measured via Borg dyspnoea and fatigue scoring). It is important to note that this is not related to the increments of daily physical activity training in the PAEP (set targets of DirectLife), which will be set by another physiotherapist through Philips website.

Statistical Analysis:

Results will be described as mean±SD or median [IQR], according to the normality in data distribution, analyzed by the Shapiro-Wilk test. In the WP1, depending on data distribution, comparisons among Actigraph GT3x and DirectLife (all the three positions) will be performed using one-way ANOVA or its correspondent Kruskal-Wallis test, with Dunn's post hoc test. To analyze DirectLife validity, correlations between PAL in both devices (week average of measured outputs in both devices) will be tested either by Pearson or Spearman correlation coefficient, depending on data distribution. To assess DirectLife's agreement with the criterion method, we will perform a Bland-Altman plot and calculate the intra-class correlation coefficient (ICC) for the energy expenditure and the time spent actively. The level of significance for all comparisons will be set at p<0.05. Data will be analyzed using the statistical package SAS version 9.3 (SAS Institute Inc, Cary, NC, USA).

For the WP2, results will be described as mean±SD or median [IQR], according to the normality in data distribution, analyzed by the Shapiro-Wilk test. Effects of the PAEP on the group of patients receiving the combined treatment (PR+PAEP) will be assessed by comparing PAL before (Visit 1) and after 3 months of the beginning of PR (Visit 2) using a paired student t-test (or the correspondent test for non-normally distributed variables). Effects of the PAEP on the main outcome (physical activity levels) will be assessed by comparing the differences (post-pre PAEP) in physical activity levels between PAEP and Control by unpaired student t-test (or the correspondent Mann-Whitney test). Correlations of PADL with other variables will be assessed either by the Pearson's or Spearman's coefficients depending on the distribution of the variables. The level of significance for all comparisons will be set at p<0.05. Data will be analyzed using the statistical package SAS version 9.3 (SAS Institute Inc, Cary, NC, USA).

Based on the study of Breyer et al. (2010) exploring the effects of a Nordic walk programme on physical activity in patients with COPD in which they show that the Nordic-walk was able to increase physical activity levels after a 3 month programme (movement intensity, 0.4+/-0.14) in comparison to controls (movement intensity, -0.05+/-0.28), for the comparison between S and C considering changes in physical activity levels as the main outcome, for an alpha of 0.05 and beta 0.1, 24 subjects are required per branch to show statistical significant differences with a 90% power. Assuming a 30% dropouts we plan to include 64 subjects (32 patients per branch, S and C).

To assess the effects of each intervention (S or C) over the short term (three months follow up period), we will perform intra-group analysis (Visit 1, Visit 2, and Visit 3), using One way ANOVA repeated measures test (or the correspondent Friedman's test for non-normally distributed variables). Effects of the PAEP on the main outcome (physical activity levels) will be assessed by comparing the differences (follow up - post PAEP, and post - pre PAEP) in physical activity levels between PAEP and Control by unpaired student t-test (or the correspondent Mann-Whitney test). Results will also be described as mean±SD or median [IQR], according to the normality in data distribution, analyzed by the Shapiro-Wilk test. Correlations of PADL with other variables will be assessed either by the Pearson's or Spearman's coefficients depending on the distribution of the variables. The level of significance for all comparisons will be set at p<0.05. Data will be analyzed using the statistical package SAS version 9.3 (SAS Institute Inc, Cary, NC, USA).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD according to Global Initiative for Chronic Obstructive Lung Disease (GOLD, 2013) referred for pulmonary rehabilitation;
* Clinical stability concerning pulmonary infections or acute exacerbations within last four weeks;
* Absence of recent Myocardial Infarction (within last 3 months), unstable angina, other significant cardiac problems, SBP > 180 mmHg, DBP > 100 mmHg or tachycardia (higher than 100 bpm);
* Absence of significant orthopaedic, neurological, cognitive and/or psychiatric impairment restricting mobility;
* Not following any exercise programme in the last 6 months.

Exclusion Criteria:

* Orthopaedic, neurological or other complaints that significantly impair normal biomechanical movement patterns, as judged by the investigator;
* Respiratory diseases other than COPD (e.g. asthma);
* COPD exacerbations within 4 weeks prior to Visit 1;
* Cognitive impairment and inability to give informed consent, as judged by the investigator;
* Involvement in the planning and/or conduct of the study;
* Participants should not be taking part in any other studies.

Ages: 30 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-02; Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Physical Activity in Daily Life (PADL) levels at 12 weeks. | 12 weeks
  The assessment of physical activity in daily life will be conducted with a validated activity monitor to assess physical activity levels (PAL) in patients with COPD, the triaxial Actigraph GT3x accelerometer. This is a small (4.6cm x 3.3cm x 1.5cm), lightweight (19 grams) and portable device that is worn around the hip to assess movement and provide several outputs reflecting PADL (i.e. raw acceleration, energy expenditure, MET rates, steps taken, physical activity intensity, subject position) by its triaxial sensor, tracking the body motion every time subjects move up, down, forwards, backwards and sideways. By measuring the acceleration of these movements, it calculates how much energy subjects used to make them. The device will be used by the patients for at least 10 hours/day during the evaluation period of one week simultaneously with the baseline assessment of PAL conducted by the DirectLife.
Change from Baseline in Physical Activity in Daily Life (PADL) levels at 24 weeks. | 24 weeks
  The assessment of physical activity in daily life will be conducted with a validated activity monitor to assess physical activity levels (PAL) in patients with COPD, the triaxial Actigraph GT3x accelerometer. This is a small (4.6cm x 3.3cm x 1.5cm), lightweight (19 grams) and portable device that is worn around the hip to assess movement and provide several outputs reflecting PADL (i.e. raw acceleration, energy expenditure, MET rates, steps taken, physical activity intensity, subject position) by its triaxial sensor, tracking the body motion every time subjects move up, down, forwards, backwards and sideways. By measuring the acceleration of these movements, it calculates how much energy subjects used to make them. The device will be used by the patients for at least 10 hours/day during the evaluation period of one week simultaneously with the baseline assessment of PAL conducted by the DirectLife.

SECONDARY OUTCOMES:
Change from Baseline in Exercise Capacity at 12 weeks. | 12 weeks
  A constant work rate test, the Endurance Shuttle Walking Test (ESWT), will be performed following an incremental shuttle walking test (ISWT). The later will assess the maximal exercise capacity of the patient and help to calculate the submaximal load (75% of the maximal load) used during the ESWT.
Change from Baseline in Exercise Capacity at 24 weeks. | 24 weeks
  A constant work rate test, the Endurance Shuttle Walking Test (ESWT), will be performed following an incremental shuttle walking test (ISWT). The later will assess the maximal exercise capacity of the patient and help to calculate the submaximal load (75% of the maximal load) used during the ESWT.
Change from Baseline in Peripheral Muscle Strength at 12 weeks. | 12 weeks
  The quadriceps maximal voluntary contraction test (QMVC) will be performed using an isokinetic machine. Patients will be sitting on a chair specifically designed to measure leg strength. Their dominant leg will be attached to a lever that will record the strength that they will produce. The test consists in measuring the strength of patients' leg applied against a steady lever. Patients will be encouraged to perform at least 3 sustained maximal knee extension of between 5 and 10 seconds duration. There will be a gap of 30-60 seconds between each contraction to allow time to recover from each effort.
  In order to assess peripheral muscle fatigue, patients will undertake a 30-repetition quadriceps contraction test using the same isokinetic machine. The test consists of 30 consecutive quadriceps contractions at 70% of patients' maximal voluntary contraction.
  All measures are very simple to perform and will be conducted after patients get familiar with the machine and the techniques.
Change from Baseline in Peripheral Muscle Strength at 24 weeks. | 24 weeks
  The quadriceps maximal voluntary contraction test (QMVC) will be performed using an isokinetic machine. Patients will be sitting on a chair specifically designed to measure leg strength. Their dominant leg will be attached to a lever that will record the strength that they will produce. The test consists in measuring the strength of patients' leg applied against a steady lever. Patients will be encouraged to perform at least 3 sustained maximal knee extension of between 5 and 10 seconds duration. There will be a gap of 30-60 seconds between each contraction to allow time to recover from each effort.
  In order to assess peripheral muscle fatigue, patients will undertake a 30-repetition quadriceps contraction test using the same isokinetic machine. The test consists of 30 consecutive quadriceps contractions at 70% of patients' maximal voluntary contraction.
  All measures are very simple to perform and will be conducted after patients get familiar with the machine and the techniques.
Change from Baseline in Health Related Quality of Life (HRQoL) at 12 weeks. | 12 weeks
  The Chronic Respiratory Questionnaire (CRQ), a specific questionnaire for patients with COPD will be applied for the assessment of the quality of life. The COPD assessment test (CAT) will also be used.
Change from Baseline in Health Related Quality of Life (HRQoL) at 24 weeks. | 24 weeks
  The Chronic Respiratory Questionnaire (CRQ), a specific questionnaire for patients with COPD will be applied for the assessment of the quality of life. The COPD assessment test (CAT) will also be used.
Change from Baseline in Acute Exacerbation rate at 12 weeks. | 12 weeks.
  Data on exacerbations that required antibiotics and/or oral corticosteroid will be recorded by asking the patients about acute exacerbations of the disease in the previous years/weeks.
Change from Baseline in Acute Exacerbations rate at 24 weeks. | 24 weeks.
  Data on exacerbations that required antibiotics and/or oral corticosteroid will be recorded by asking the patients about acute exacerbations of the disease in the previous years/weeks.
Change from Baseline in Degree of Dyspnoea at 12 weeks. | 12 weeks
  The Medical Research Council Scale (MRC) will be used to evaluate the sensation of dyspnoea during daily living activities.
Change from Baseline in Degree of Dyspnoea at 24 weeks. | 24 weeks
  The Medical Research Council Scale (MRC) will be used to evaluate the sensation of dyspnoea during daily living activities.
Change from Baseline in Anxiety and Depression levels at 12 weeks. | 12 weeks
  Levels of anxiety and depression will be measured by the Hospital Anxiety and Depression Scale (HADS).
Change from Baseline in Anxiety and Depression levels at 24 weeks. | 24 weeks
  Levels of anxiety and depression will be measured by the Hospital Anxiety and Depression Scale (HADS).
Change from Baseline in psychological status at 12 weeks | 12 weeks
  A number of psychological constructs will be measured using a number or different (validated) questionnaires. The constructs we are measuring are: Coping with problems¬, positive health (psychosocial wellbeing), social support, self-efficacy, affect, and motivation.
Change from Baseline in psychological status at 24 weeks | 24 weeks
  A number of psychological constructs will be measured using a number or different (validated) questionnaires. The constructs we are measuring are: Coping with problems¬, positive health (psychosocial wellbeing), social support, self-efficacy, affect, and motivation.
Change from Baseline in Systemic inflammation at 12 weeks | 12 weeks
  Levels of systemic inflammation (White blood cells, serum C-reactive protein and circulating cytokines) will be assessed in blood samples. Twenty milliliters (20 ml) of blood will be obtained in a serum tube (brown). Spin at 1200 rpm. Serum aliquot and stored at -80 degree. Samples will be identified with the date and the patients' study id (anonymised id). Serum C-reactive protein (CRP) concentrations will be measured using a highly sensitive immunonephelometric assay. Serum cytokine assessment will be carried out using Cytometric Bead Array (CBA) for simultaneous detection of ten cytokines in serum.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Rabinovich, Post PhD, Principal Investigator — University of Edinburgh
Locations (1):
- Physiotherapy Department - Leith Community Treatment Centre, Edinburgh, United Kingdom

REFERENCES:
- [Background] Pitta F, Troosters T, Spruit MA, Probst VS, Decramer M, Gosselink R. Characteristics of physical activities in daily life in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 May 1;171(9):972-7. doi: 10.1164/rccm.200407-855OC. Epub 2005 Jan 21. PMID 15665324
- [Background] Garcia-Aymerich J, Lange P, Benet M, Schnohr P, Anto JM. Regular physical activity reduces hospital admission and mortality in chronic obstructive pulmonary disease: a population based cohort study. Thorax. 2006 Sep;61(9):772-8. doi: 10.1136/thx.2006.060145. Epub 2006 May 31. PMID 16738033
- [Background] Nici L, Donner C, Wouters E, Zuwallack R, Ambrosino N, Bourbeau J, Carone M, Celli B, Engelen M, Fahy B, Garvey C, Goldstein R, Gosselink R, Lareau S, MacIntyre N, Maltais F, Morgan M, O'Donnell D, Prefault C, Reardon J, Rochester C, Schols A, Singh S, Troosters T; ATS/ERS Pulmonary Rehabilitation Writing Committee. American Thoracic Society/European Respiratory Society statement on pulmonary rehabilitation. Am J Respir Crit Care Med. 2006 Jun 15;173(12):1390-413. doi: 10.1164/rccm.200508-1211ST. No abstract available. PMID 16760357
- [Background] Pitta F, Troosters T, Probst VS, Langer D, Decramer M, Gosselink R. Are patients with COPD more active after pulmonary rehabilitation? Chest. 2008 Aug;134(2):273-280. doi: 10.1378/chest.07-2655. Epub 2008 Apr 10. PMID 18403667
- [Background] Breyer MK, Breyer-Kohansal R, Funk GC, Dornhofer N, Spruit MA, Wouters EF, Burghuber OC, Hartl S. Nordic walking improves daily physical activities in COPD: a randomised controlled trial. Respir Res. 2010 Aug 22;11(1):112. doi: 10.1186/1465-9921-11-112. PMID 20727209
- [Background] de Blok BM, de Greef MH, ten Hacken NH, Sprenger SR, Postema K, Wempe JB. The effects of a lifestyle physical activity counseling program with feedback of a pedometer during pulmonary rehabilitation in patients with COPD: a pilot study. Patient Educ Couns. 2006 Apr;61(1):48-55. doi: 10.1016/j.pec.2005.02.005. Epub 2006 Feb 7. PMID 16455222
- [Background] Rabinovich RA, Louvaris Z, Raste Y, Langer D, Van Remoortel H, Giavedoni S, Burtin C, Regueiro EM, Vogiatzis I, Hopkinson NS, Polkey MI, Wilson FJ, Macnee W, Westerterp KR, Troosters T; PROactive Consortium. Validity of physical activity monitors during daily life in patients with COPD. Eur Respir J. 2013 Nov;42(5):1205-15. doi: 10.1183/09031936.00134312. Epub 2013 Feb 8. PMID 23397303
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278